CLINICAL TRIAL: NCT01667198
Title: Quality Improvement in Screening Colonoscopy - a Randomized Trial of Tailored Training Intervention Versus Simple Feedback on the Quality Indicators.
Brief Title: Randomized Study of Train the Colonoscopy Leaders Course Versus Audit and Feedback on Colonoscopy Quality Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); University of Oslo (Other); Erasmus Medical Center (Other); Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IP2010016270
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Train the leaders course (Experimental)
  Interventions: Procedure: Train the leaders course
- Audit and feedback (Active Comparator)
  Interventions: Behavioral: Audit and feedback

INTERVENTIONS:
Procedure: Train the leaders course — Screening centre leaders randomized to the training intervention group will be invited to take part in a train-the-leaders course. The Train-the-leaders course will consist of three phases: (i) pre-training assessment, (ii) hands-on-training and (iii) post-training evaluation and feedback. The Train-the-leaders course will be run in polish by the team from the Maria Sklodowska-Curie Memorial Cancer Center and Institute on Oncology, Warsaw, which was trained in delivering such intervention by experts from the United Kingdom.
  Arms: Train the leaders course
Behavioral: Audit and feedback — Screening centre leaders randomized to the feedback group will receive (by e-mail and conventional mail) feedback on their individual screening colonoscopy quality indicators (adenoma detection rate and ceacal intubation rate) measured for the 2011 edition of the national screening program. The results will be presented in a league table in order to enable comparison with anonymous results of all endoscopists who performed at least 30 colonoscopies within the screening program. In addition, a link to a webpage containing data on individual and overall colonoscopy quality indicators over the last four years of the screening program will be provided.
  Arms: Audit and feedback

SUMMARY:
Professional societies recommend that endoscopists measure their ceacal intubation rate, adenoma detection rate as indicators of the screening colonoscopy quality. However, it is uncertain how to improve adenoma detection rate and reduce inter-endoscopists' variability in the detection of adenomas. The investigators hypothesize that a hands-on-training intervention tailored to the results of environmental assessment and audit on colonoscopy quality indicators results in higher adenoma detection rate improvement than simple audit and feedback. The investigators further hypothesize that by training the leaders of the screening centres, the effect of the intervention will be further disseminated among other endoscopists from the participating centers, and will thus result in additional increase in individual adenoma detection rate.

The primary aim is to compare the impact on adenoma detection rate of two screening colonoscopy improvement programs:

1. Tailored training intervention.
2. Audit feedback on colonoscopy quality indicators.

ELIGIBILITY:
Inclusion Criteria:

* screening center leading colonoscopist
* at least 30 screening colonoscopies in the 2011 edition of the screening program
* adenoma detection rate lower than 25%

Exclusion Criteria:

* lack of participation in the 2012 edition of the screening program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Screening centre leader's adenoma detection rate | till the end of calendar year after the training intervention
  Adenoma detection rate is defined as the proportion of screened subjects in whom at least one adenomatous lesion is identified.

SECONDARY OUTCOMES:
Screening center's overall adenoma detection rate | Till the end of calendar year after the training intervention
  Adenoma detection rate is defined as the proportion of screened subjects in whom at least one adenomatous lesion is identified.
Screening centre leader's proximal and distal adenoma detection rate | Till the end of calendar year after the training intervention
  Adenoma detection rate is defined as the proportion of screened subjects in whom at least one adenomatous lesion is identified.
Screening centre's non-polypoid lesion detection rate | Till the end of calendar year after the training intervention
Overall screening centre's ceacal intubation rate | Till the end of calendar year after the training intervention
  Ceacal intubation is defined as the passage of the colonoscope tip to a point proximal to the ileoceacal valve and visualization of the entire ceacum.
Screening centre leader's withdrawal technique | Till the end of calendar year after the training intervention
  Withdrawal technique assessed by a trained endoscopy nurse

CONTACTS AND LOCATIONS:
Overall Officials: Michal F. Kaminski, MD, PhD, Principal Investigator — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology; Jaroslaw Regula, MD, PhD, Study Chair — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
Locations (1):
- The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland

REFERENCES:
- [Derived] Kaminski MF, Anderson J, Valori R, Kraszewska E, Rupinski M, Pachlewski J, Wronska E, Bretthauer M, Thomas-Gibson S, Kuipers EJ, Regula J. Leadership training to improve adenoma detection rate in screening colonoscopy: a randomised trial. Gut. 2016 Apr;65(4):616-24. doi: 10.1136/gutjnl-2014-307503. Epub 2015 Feb 10. PMID 25670810